CLINICAL TRIAL: NCT06410105
Title: Three-dimensional Assessment of Root Resorption Following Treatment With Clear Aligners Using Cone Beam Computed Tomography
Brief Title: Orthodontic Treatment With Clear Aligner
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tishreen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Tishreen U _orthodontic
Record Dates: First submitted 2024-05-04; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2020-12

CONDITIONS: Orthodontic Pathological Resorption of External Root
Keywords: Orthodontic, clear aligners, fixed appliances, CBCT

STUDY DESIGN:
Intervention Model Description: : Crossover Assignment A randomized, controlled, crossover, double-blind clinical study, Comparison of
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Groub(1): 13 patient treated with CLEAR ALIGNERS (Experimental): The CA group included 13 patients treated with clear aligners Tree-dimensional images were captured using a CBCT scan (KaVo® Dental GmbH, Bismarckring, Germany). Te pre-treatment imaging parameters were 120 kV, 5 mA, 0.3 mm voxel size, and a feld of view of 230×170 mm
  Interventions: Device: CLEAR ALIGNERS
- Groub(2): 13 patient treated with a fixed orthodontic (Experimental): . The FA group included 13 patients treated with a fxed orthodontic appliance (american orthodontics, WI.Sheboygam, USA). Tree-dimensional images were captured using a CBCT scan (KaVo® Dental GmbH, Bismarckring, Germany). Te pre-treatment imaging parameters were 120 kV, 5 mA, 0.3 mm voxel size, and a feld of view of 230×170 mm, which
  Interventions: Device: CLEAR ALIGNERS

INTERVENTIONS:
Device: CLEAR ALIGNERS — The CA group included 13 patients treated with clear aligners Tree-dimensional images were captured using a CBCT scan (KaVo® Dental GmbH, Bismarckring, Germany). Te pre-treatment imaging parameters were 120 kV, 5 mA, 0.3 mm voxel size, and a feld of view of 230×170 mm

SUMMARY:
Three-dimensional Assessment of Root Resorption following treatment with clear aligners using Cone Beam Computed Tomography Design: A randomized, controlled, crossover, double-blind clinical study including twenty six adult , aged 18-25 years old.

DETAILED DESCRIPTION:
Orthodontically induced root resorption is one of the common undesirable sequalae of orthodontic treatment. one third of the patients treated with fixed appliances showed more than 3 mm of root resorption whereas at least 2% of orthodontic patients showed more than 5 mm of root resorption.

There is a controversy in the literature regarding the effect of clear aligners on apical root resorption. One previous study reported that some kinds of removable aligners may have the potential of minimizing orthodontic ally induced root resorption due to the studied piezoelectric property by these materials Till now, the degree of apical root resorption following treatment with (in house) aligners has not been reported in the literature.

ELIGIBILITY:
Inclusion Criteria:

The Clinical Diagnosis the age of patients ranges between 18-25 years, medium crowding between 3-6 mm in the area of the upper anterior teeth according to Little irregularity index 20,class1 according angel classification healthy patient No previous orthodontic treatment vital teeth with periodontal tissue without root absorption,

Exclusion Criteria:

Previous history of orthodontic or orthopedic treatment. Presence of craniofacial anomalies. Presence of any signs and symptoms of gingival and periodontal diseases. Presence of significant medical history (including drug allergy). Pregnant and lactating women

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2020-12-19 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
treatment with clear aligners | two years
  to determine the root resorption for upper anterior teeth following treatment with clear aligners orthodontic appliances CA comparison with fixed appliances using CBCT.)

SECONDARY OUTCOMES:
comparative study of Buccolingual Inclination changes | two years
  to evaluate the Buccolingual Inclination changes and for upper anterior teeth following treatment with clear aligners orthodontic appliances CA comparison with fixed appliances using CBCT.

CONTACTS AND LOCATIONS:
Overall Officials: fadi khalil, prof, Study Chair — Tishreen University
Locations (1):
- Tishreen University, Latakia, Syria

IPD SHARING:
Plan to Share IPD: Yes
study protocol ,Informed Consent From
Supporting Information: ICF
Time Frame: 9 month